CLINICAL TRIAL: NCT07079306
Title: Engagement and Satisfaction With a ChatGPT-Supported Text Messaging Program for Smoking Cessation
Brief Title: ChatGPT-Supported Text Messaging Program for Smoking Cessation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GWUniversity
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; ai; text messaging
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Text messages about quitting smoking and access to specialized ChatGPT chatbot
  Interventions: Behavioral: BeFree+Bot
- Control (Active Comparator): Text messages about quitting smoking
  Interventions: Behavioral: BeFree

INTERVENTIONS:
Behavioral: BeFree+Bot — Text messaging program called BeFree and access to BBot, ChatGPT chatbot
  Arms: Intervention
Behavioral: BeFree — Text messaging program called BeFree
  Arms: Control

SUMMARY:
The current research proposal aims to explore how a purpose driven LLM ChatGPT chatbot, BeFreeBot, might enhance an evidence-based text messaging smoking cessation program, BeFree. The research will consist of a formative evaluation comparing quitting related outcomes among users of BeFree+Bot and BeFree.

ELIGIBILITY:
Inclusion Criteria:

* lives in the US
* smoked a cigarette within the last 7 days
* has a mobile phone
* willing to receive text messages about the health effects of smoking on their mobile phone for 30 days

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Continuous abstinence | at 1 month follow-up
  the longest continuous period (in days) that you did not smoke a cigarette

CONTACTS AND LOCATIONS:
Locations (1):
- Prolific, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
It is a small pilot study